CLINICAL TRIAL: NCT06265623
Title: Prospective Observational Study to Assess the Influence of Intermittent Hypoxaemia on Lung Function Decline, Morbidity, and Mortality in COPD Patients (PROSA Study)
Brief Title: Intermittent Hypoxemia, Lung Function Decline, Morbidity, and Mortality in COPD (PROSA Study).
Acronym: PROSA
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Rainer H. Böger, Prof. Dr. med. Dr. h.c., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: UKE-IKPT 2024/01
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: lung function, prognosis, exercise testing, spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for plasma biomarker analysis and DNA extraction for genotyping of single nucleotide polymorphisms in target genes of the L-arginine-dimethylarginine-NO pathway.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients with exertional desaturation: Patients with chronic obstructive pulmonary disease stages 2-3, groups B or E according to the GOLD Guideline (2023), who experience a drop in arterial oxygen saturation (by pulse oximetry) to <90% or a drop by 4% or greater of the basal value during a six-minute walk test.
  Interventions: Other: No active intervention, but observational follow-up
- COPD patients without exertional desaturation: Patients with chronic obstructive pulmonary disease stages 2-3, groups B or E according to the GOLD Guideline (2023), who do not experience a drop in arterial oxygen saturation (by pulse oximetry) to <90% or a drop by 4% or greater of the basal value during a six-minute walk test.
  Interventions: Other: No active intervention, but observational follow-up

INTERVENTIONS:
Other: No active intervention, but observational follow-up — Patients remain in usual care by their pulmonary medicine specialists and are being observed during annual follow-up investigations during up to 3 years

SUMMARY:
This study aims to analyze if patients with chronic obstructive lung disease who experience a decline of blood oxygen saturation during physical exercise have a disease course different from that of COPD patients who do not experience a decline in blood oxygen saturation during exercise. Patients will be followed for a total of 3 years.

DETAILED DESCRIPTION:
The major aim of the study is to test whether intermittent hypoxaemia is a major driver of the progression of chronic obstructive lung disease (COPD). The second aim is to analyse whether dysregulation of the L-arginine / dimethylarginine pathway is a mechanistic link between intermittent hypoxemia and lung function decline, and whether plasma biomarkers are suitable to identify COPD patients at high risk of rapid lung function decline and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes with a diagnosis of chronic obstructive lung disease (COPD) stages 2-3, groups B and E according to GOLD 38 as assessed by their primary family doctor or pneumology specialist who are treated with long-acting bronchodilators on a stable dose for at least four months prior to inclusion into the study;
2. Age at inclusion 18 - 80 years;
3. Physical ability and willingness to perform 6-minute walk testing and bicycle ergometry testing;
4. Signed written informed consent form

Exclusion Criteria:

1. Participation in another clinical study within the last 3 months before inclusion into the present study;
2. Any somatic or psychic disease that may hamper participation in the study or compliance with the study protocol (at the investigator's discretion);
3. Any somatic disease that puts the patient at increased risk when performing the exercise tests or impairs the patient's ability to properly perform the exercise tests, like advanced coronary artery disease, advanced chronic heart failure, uncontrolled hypertension, orthopaedic, or neurological diseases (non-exclusive list of examples);
4. Any disease or health condition that reduces the patient's life expectancy to less than the expected time frame of this study, other than chronic obstructive lung disease (at the investigator's discretion);
5. Pregnancy or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted a patients with chronic obstructive pulmonary disease of all sexes aged 18 - 80 years. They must be graded as stage 2 - 3 according to GOLD criteria (FEV1 between 30 and 79% of the age-adjusted predicted value) and belong to groups B or E according to symptom scores (mMRC or CAT questionnaires) and exacerbation history.
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in FEV1(% of LLN) between baseline and end-of-follow-up | 3 years
  The difference in measured FEV1 assessed by spirometry and expressed as percent of the lower limit of the normal distribution based upon the Global Lung Function 2022 Equations, by comparing results of the baseline measurement with those of the last investigation during up to three years of follow-up

SECONDARY OUTCOMES:
Difference in all-cause mortality during follow-up between groups | 3 years
  Number of patients who died from any cause during follow-up in either of the two groups.
Difference in COPD-related mortality during follow-up between groups | 3 years
  Number of patients who died from COPD and its complications during follow-up in either of the two groups.
Difference in frequency of hospital admissions for exacerbation of COPD during follow-up between groups | 3 years
  Number of patients who were admitted to hospital because of exacerbated COPD during follow-up in either of the two groups.
Difference in frequency of hospital admissions for causes other than exacerbation of COPD during follow-up between groups | 3 years
  Number of patients who were admitted to hospital for any other reason than exacerbated COPD during follow-up in either of the two groups.
Sensitivity of plasma biomarkers (spec. ADMA and SDMA) to predict the prevalence of exertional desaturation in COPD patients | 3 years
  Sensitivity analysis (ROC analysis) of biomarkers and presence of exertional desaturation (as defined in the protocol) or not in study participants.
Sensitivity and specificity of plasma biomarkers (spec. ADMA and SDMA) measured at baseline to prospectively predict the slope of lung function decline in COPD patients | 3 years
  Prospective survival analysis (Kaplan-Meier) of plasma biomarkers measured at the time of study inclusion and the difference in FEV1(% of lower limit of normal) between baseline and last measurement during follow-up.
Sensitivity and specificity of plasma biomarkers at baseline to prospectively predict the mortality rate in COPD patients | 3 years
  Prospective survival analysis (Kaplan-Meier) of plasma biomarkers measured at the time of study inclusion and total mortality during follow-up.
Difference in incidence and extent of exercise hypoxemia between carriers and non-carriers of single nucleotide polymorphisms (SNPs) in genes of the L-arginine - dimethylarginine pathway | 3 years
  Comparison of the rates of prevalence of exertional desaturation between homozygous carriers of the major versus minor allele of SNPs in the NOS III, DDAH1, DDAH2, PRMT1-9, AGXT2, and ARG1-2 genes.
Difference in positive and negative predictive value of bicycle ergometry, 6-minute walk test, and 15-sec breath-hold test to discriminate between COPD patients with exertional desaturation versus those without exertional desaturation | 3 years
  Comparison of sensitivity and specificity analyses (ROC analyses) of the outcome of named exercise tests to detect exertional desaturation in study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Böger, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Institute of Clinical Pharmacology and Toxicology, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable individual request, IPD can be made available for further analyses by other researchers.
Supporting Information: Study Protocol
Time Frame: Data can be made available after conclusion of the trial and final analysis.
Access Criteria: Written, reasoned request to either of the two principal contact persons of the study.

REFERENCES:
- [Derived] Boger R, Hannemann J. Defining the role of exertional hypoxemia and pulmonary vasoconstriction on lung function decline, morbidity, and mortality in patients with chronic obstructive lung disease - the PROSA study: rationale and study design. BMC Pulm Med. 2024 May 30;24(1):262. doi: 10.1186/s12890-024-03074-x. PMID 38816826